CLINICAL TRIAL: NCT07046364
Title: The Effect of Remimazolam on Emergence Delirium in Pediatrics Undergoing Neurosurgery With Sevoflurane Anesthesia
Brief Title: Remimazolam and Emergence Delirium in Pediatrics
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Mu Dong Liang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-407-002
Record Dates: First submitted 2025-06-15; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-12

CONDITIONS: Pediatric; Neurosurgery; Sevoflurane Anesthesia; Remimazolam; Emergence Delirium
Keywords: emergence delirium; remimazolam; pediatric; neurosurgery; sevoflurane anesthesia
MeSH Terms: conditions — Emergence Delirium | interventions — remimazolam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam group (Experimental): A loading dose of remimazolam 0.3 mg/Kg was given at anesthesia induction and followed with 1 mg/Kg/h until 10 minutes before the end of surgery. Sevoflurane was used to maintain BIS between 40-60.
  Interventions: Drug: Remimazolam
- Normal saline group (Placebo Comparator): An identical volume of normal saline was given as placebo. Patients received sevoflurane to maintain anesthesia depth (BIS) 40-60
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Remimazolam — After anesthesia induction, a loading investigational drug at a rate of [3.6*kg] ml/h (lasting for 5 minutes, equivalent to 0.3 mg/kg of remimazolam), and then adjust the infusion rate to [1*kg] ml/h (equivalent to 1 mg/kg of remimazolam). The infusion is expected to stop 10 minutes before the end of the surgery.
  Arms: Remimazolam group
Drug: Normal Saline — After anesthesia induction, a loading investigational drug at a rate of [3.6*kg] ml/h (lasting for 5 minutes, equivalent to 0.3 mg/kg of normal saline), and then adjust the infusion rate to [1*kg] ml/h (equivalent to 1 mg/kg of normal saline). The infusion is expected to stop 10 minutes before the end of the surgery.
  Arms: Normal saline group

SUMMARY:
Emergence delirium is a common complication in pediatrics undergoing neurosurgery. Previous study showed that a single bolus of remimazolam was associated with lower incidence of postoperative agitation. Present study was designed to investigate if remimazolam supplemented to sevoflurane anesthesia could decrease the risk of emergence delirium in pediatrics undergoing neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 to 6 years old
* Planned to receive elective neurosurgery under general anesthesia
* Expected duration of surgery > 1 hour

Exclusion Criteria:

* Allergy to benzodiazepine
* Use of other sedatives within 12 hours before surgery such as benzodiazepines, propofol, chloral hydrate, etc.,
* ASA classification IV or above
* Unable to complete emergence delirium assessment, such as language, hearing or vision impairment.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 248 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Emergence delirium | The subjects were evaluated at 10 minutes, 20 minutes, 30 minutes after admission to PACU or before discharge
  The Cornell Assessment of Pediatric Delirium (CAPD) was used to assess delirium. It consists of a total of 8 items, with each item scored from 0 to 4. Delirium can be diagnosed when the total score is ≥ 10.

SECONDARY OUTCOMES:
Postoperative delirium | Delirium was assessed at 07:00~09:00 and 17:00~20:00 on the 1st, 2nd and 3rd day after surgery
  The Cornell Assessment of Pediatric Delirium (CAPD) scale was used to assess whether the subjects developed delirium. It consists of a total of 8 items, with each item scored from 0 to 4. Delirium can be diagnosed when the total score is ≥ 10.
Pain score | Pain intensity was assessed at 07:00~09:00 and 17:00~20:00 on the 1st, 2nd and 3rd day after surgery
  The FLACC behavioral rating scale was used to evaluate the pain intensity. It mainly includes five indicators: Facial Expression, Legs, Activity, Cry, and Consolability. The score is the sum of the above five indicators, ranging from a minimum of 0 to a maximum of 10. A higher score indicates more obvious discomfort and pain.
Sleep quality within 3 days after surgery | Within 3 days after surgery
  The Numeric Rating Scale (NRS) was used for sleep quality assessment of children by their parents/caregivers within 3 days after surgery. The scores of NRS ranging from a minimum of 0 to a maximum of 10. A lower score indicates poorer sleep quality.
Sleep quality 7 days after surgery and 1 month after surgery | 7 days after surgery and 1 month after surgery
  The Tayside Children's Sleep Questionnaire (TCSQ) was adopted to assess the sleep quality 7 days after surgery and 1 month after surgery.The TCSQ consists of 10 questions, with scores ranging from a minimum of 0 to a maximum of 40. A higher score indicates poorer sleep quality.
Postoperative adverse behavior change | 1st, 3rd days after surgery
  Post-hospitalization behavior questionnaire (PHBQ) was used to evaluate the postoperative adverse behavior change. It consists of 26 items, with scores ranging from a minimum of -52 to a maximum of 52. A higher score indicates poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No